CLINICAL TRIAL: NCT04587297
Title: Food Collection From Type 1 Diabetic Patients Practicing Insulin Functional Therapy : GLUCAL2
Brief Title: Food Collection From Type 1 Diabetic Patients Practicing Insulin Functional Therapy
Acronym: GLUCAL2
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0552
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Type 1
Keywords: Diabetes; Functional insulin therapy; carbohydrate counting
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
a food collection will be performed in this study with type 1 diabetic patients trained to carbohydrate counting, to collect data on the meals consumed daily and their quantities for a period of 1 month.

ELIGIBILITY:
Inclusion criteria:

* type 1 diabetic patients
* Using carbohydrate counting and functional insulin therapy
* Patient with Social security or beneficiary
* Patient able to read and understand the procedure, and able to express consent for the study protocol

Exclusion criteria:

* Patient abusing substances
* person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure -- Patient having a psychological conditions making him unable to follow and understand study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
number of meals | one month
  our primary outcome is to collect the description of 2000 meals from different patients correctly described.

CONTACTS AND LOCATIONS:
Overall Officials: Eric RENARD, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC